CLINICAL TRIAL: NCT00573976
Title: United States Multi-Center Study to Assess the Validity and Reliability of the Spinal Cord Independence Measure (SCIM III)
Brief Title: Study to Assess the Validity and Reliability of the Spinal Cord Independence Measure (SCIM III)
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: University of Pittsburgh (Other); University of Texas Southwestern Medical Center (Other); Rancho Los Amigos National Rehabilitation Center (Other); University of Missouri-Columbia (Other); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); VA Long Beach Healthcare System (U.S. Federal Agency); Allina Health System (Other); University of Kentucky (Other); Mayo Clinic (Other); University of Louisville (Other); Shirley Ryan AbilityLab (Other); Wake Forest University Health Sciences (Other); Kessler Foundation (Other); MedStar National Rehabilitation Network (Other); MetroHealth Rehabilitation Institute of Ohio (Unknown); Touro Rehabilitation Center (Unknown); Icahn School of Medicine at Mount Sinai (Other); Medical College of Wisconsin (Other); Unity Health Toronto (Other); Thomas Jefferson University (Other); The Institute for Rehabilitaion and Research Foundation (Other)
Responsible Party: Kimberly D. Anderson, Ph.D, University of California, Irvine
Other Study IDs: OCRT07019; 2007-5854
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Spinal Cord Injury
Keywords: SCIM; SCIM III; Multi-Center; United States
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the past two decades there have been great strides made in understanding the biological changes resulting from spinal cord injury (SCI). The future holds promise of the development of therapies that will promote degrees of repair and recovery of function for people living with SCI. Lessons learned from past "failed" SCI clinical trials, however, demonstrate that, in order to accurately evaluate the overall effectiveness of SCI therapies, more sensitive outcomes measures are needed. Specifically, and reflecting the ultimate goal of clinical interventions - inducing functional recovery - the Spinal Cord Independence Measure (SCIM), has been recommended for further testing and development for use as a measure of functional ability in future SCI clinical studies. The SCIM is a very simple questionnaire and score sheet that an evaluator uses to determine how independently a person with SCI can perform certain tasks.

A panel of SCI researchers recommended the SCIM as the most suitable among four candidate measures of functional recovery reviewed at a special meeting sponsored by the National Institute on Disability and Rehabilitation Research (NIDRR) at a joint meeting of the American Spinal Injury Association and the International Spinal Cord Society (ASIA-ISCoS) in Boston, MA, in June 2006. It was recommended that a large-scale, multi-center, prospective trial be conducted in the United States, which would mirror a recently published multi-site international study.

The proposed research on the SCIM III, the latest and most sensitive version of the SCIM, would test the hypothesis that the SCIM III is a valid, reliable, and sensitive measure of functional ability in persons with SCI. Twenty-two rehabilitation centers throughout the United States will enroll a maximum of 660 subjects. Functional ability will be measured with the SCIM III during the first week of admittance into inpatient acute rehabilitation and within one week of discharge from the same rehabilitation program. Statistical analyses will be used to test the validity, reliability, and sensitivity of the SCIM III. The results will demonstrate whether the SCIM III is a suitable outcome measure to assess SCI specific functional ability in future clinical trials.

DETAILED DESCRIPTION:
STUDY PURPOSE This clinical research study will be performed to assess the validity, reliability, and sensitivity of the Spinal Cord Independence Measure (SCIM III) in measuring functional ability in persons with spinal cord injury (SCI).

Aims and Hypothesis:

Overall hypothesis - The SCIM III is a valid, reliable, and sensitive measure of functional ability in persons with SCI.

Aim 1: Examine the validity of the SCIM III as an outcome measure to assess functional ability in persons with SCI.

1. Criterion-related validity
2. Construct validity of components

Aim 2: Examine the reliability of SCIM III evaluations.

1. Inter-rater reliability
2. Internal consistency

Aim 3: Examine the sensitivity of the SCIM III to functional change.

1. Sensitivity to functional change compared to the Functional Independence Measure (FIM).
2. Sensitivity to functional change over time

STUDY DESIGN This is a multi-center, prospective clinical research study performed to assess the validity, reliability, and sensitivity of the Spinal Cord Independence Measure (SCIM III) in measuring functional ability in persons with spinal cord injury (SCI).

UCI will act as the coordinating center for this study, collecting and performing statistical data analysis. There will be approximately 22 rehabilitation centers participating in this study. De-identified data will be transferred from these sites to Dr. Kim Anderson at UCI.

ELIGIBILITY:
Inclusion Criteria:

* Any level SCI
* Traumatic or non-traumatic cause of spinal injury
* ASIA Impairment Scale grade A, B, C, or D
* Males and females 18 years of age or older

Exclusion Criteria:

* Cognitive impairments
* Any additional condition, other than SCI and SCI-related secondary conditions, that may influence everyday function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The characteristics of the proposed subject population include:
  * Males and females 18 years of age or older
  * Adults who are competent to give informed consent
  * Subjects who are able to read or speak English
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2007-09; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly D Anderson, Ph.D., Principal Investigator — University of California, Irvine